CLINICAL TRIAL: NCT03577093
Title: Study on the Molecular Mechanism of miR-494 Mediating Cell Cycle Regulation Following Cerebral Ischemia
Brief Title: Molecular Mechanisms of microRNA-494 Involving in Cerebral Ischemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Vice President of Xuanwu Hospital,Capital Medical University, Capital Medical University
Other Study IDs: miR-494
Record Dates: First submitted 2018-06-22; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Ischemic Stroke
Keywords: stroke, miR-494, neuroprotection, CDK
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ischemic stroke: acute ischemic stroke patients within 6h after stroke onset
  Interventions: Other: There is no intervention at all.
- control: healthy controls
  Interventions: Other: There is no intervention at all.

INTERVENTIONS:
Other: There is no intervention at all. — There is no intervention at all.

SUMMARY:
We and other investigations suggested that the activation of nerve cell cycle following cerebral ischemia led to neuronal apoptosis, glial cell proliferation and the formation of glial scar.The cyclin-dependent kinases (CDKs) and cyclins jointly promoted the cell cycle progression. Our preliminary clinical trial found a new microRNA-miR-494, which involved in the occurrence of acute ischemic stroke. In our animal experiment, miR-494 could relieve cerebral ischemia injury through inhibiting cyclin-dependent kinase 6(CDK6), ubiquitin-conjugating enzyme E2L6 (UBE2L6) and histone deacetylase 3 (HDAC3), which suggested that miR-494 might play an important role in the regulation of cell cycle following cerebral ischemia. This project intends to verify the following hypothesis：①miR-494 suppresses CDK6, and/or fibroblast growth factor16(FGF16)-Ras-extracellular signal-regulated kinase(ERK)--v-myc avian myelocytomatosis viral oncogene homolog(MYC) pathway, and/or phosphatase and tensin homolog(PTEN)-/protein kinase B(AKT)-mechanistic target of rapamycin(mTOR)-S6k pathway;②miR-494 inhibits UBE2L6, upregulates the hypoxia-inducible factor 1 α(HIF-1α) expression in nerve cells, thereby increases the p21 and p27 protein levels and inhibits cyclin-dependent kinase2(CDK2)activity;③miR-494 represses HDAC3 and downregulates the cyclin-dependent kinase1(CDK1)protein level. These all mediate the cell cycle arrest of neurons and astrocytes, reduce the neuronal apoptosis and glial scar formation,promote the recovery of neurological function and provide new targets for the treatment of ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* (1）diagnosis of first ischemic stroke based on clinical information and magnetic resonance imaging; (2)presentation of subjects within 6h of the event; (3)National Institutes of Health Stroke Scale (NIHSS) score between 4 and 15.

Exclusion Criteria:

* (1）suspected cardiogenic embolism;(2）secondary stroke from cerebral hemorrhage, trauma, cancer or aneurysm and so on;(3）bleeding tendency;(4）severe cardiac,pulmonary,hepatic or renal insufficiency;(5）Vital signs are unstable to be assessed.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: acute ischemic stroke patients who were presented within 6h of the event would be recruited to this study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-06-06 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
the molecular mechanism of miR-494 mediating cell cycle regulation following cerebral ischemia | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Luo Yumin, Principal Investigator — Capital Medical University
Locations (1):
- Xuanwu Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for all primary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent panel.Requestors will be required to sign a Data Access Agreement.
URL: http://bethesda.org

REFERENCES:
- [Background] Bizen N, Inoue T, Shimizu T, Tabu K, Kagawa T, Taga T. A growth-promoting signaling component cyclin D1 in neural stem cells has antiastrogliogenic function to execute self-renewal. Stem Cells. 2014 Jun;32(6):1602-15. doi: 10.1002/stem.1613. PMID 24302516
- [Background] Zhao H, Wang J, Gao L, Wang R, Liu X, Gao Z, Tao Z, Xu C, Song J, Ji X, Luo Y. MiRNA-424 protects against permanent focal cerebral ischemia injury in mice involving suppressing microglia activation. Stroke. 2013 Jun;44(6):1706-13. doi: 10.1161/STROKEAHA.111.000504. Epub 2013 Apr 23. PMID 23613494
- [Result] Iyirhiaro GO, Zhang Y, Estey C, O'Hare MJ, Safarpour F, Parsanejad M, Wang S, Abdel-Messih E, Callaghan SM, During MJ, Slack RS, Park DS. Regulation of ischemic neuronal death by E2F4-p130 protein complexes. J Biol Chem. 2014 Jun 27;289(26):18202-13. doi: 10.1074/jbc.M114.574145. Epub 2014 May 14. PMID 24828495
- [Result] Nobs L, Baranek C, Nestel S, Kulik A, Kapfhammer J, Nitsch C, Atanasoski S. Stage-specific requirement for cyclin D1 in glial progenitor cells of the cerebral cortex. Glia. 2014 May;62(5):829-39. doi: 10.1002/glia.22646. Epub 2014 Feb 19. PMID 24550001
- [Result] Demyanenko S, Uzdensky A. Profiling of Signaling Proteins in Penumbra After Focal Photothrombotic Infarct in the Rat Brain Cortex. Mol Neurobiol. 2017 Nov;54(9):6839-6856. doi: 10.1007/s12035-016-0191-x. Epub 2016 Oct 22. PMID 27771897
- [Result] Zhao H, Luo Y, Liu X, Wang R, Yan F, Liu X, Li S, Leak RK, Ji X. Ischemic post-conditioning partially reverses cell cycle reactivity following ischemia/reperfusion injury: a genome-wide survey. CNS Neurol Disord Drug Targets. 2013 May 1;12(3):350-9. doi: 10.2174/1871527311312030008. PMID 23469856
- [Result] Liu L, Lu Y, Martinez J, Bi Y, Lian G, Wang T, Milasta S, Wang J, Yang M, Liu G, Green DR, Wang R. Proinflammatory signal suppresses proliferation and shifts macrophage metabolism from Myc-dependent to HIF1alpha-dependent. Proc Natl Acad Sci U S A. 2016 Feb 9;113(6):1564-9. doi: 10.1073/pnas.1518000113. Epub 2016 Jan 25. PMID 26811453
- [Result] Fournier M, Orpinell M, Grauffel C, Scheer E, Garnier JM, Ye T, Chavant V, Joint M, Esashi F, Dejaegere A, Gonczy P, Tora L. KAT2A/KAT2B-targeted acetylome reveals a role for PLK4 acetylation in preventing centrosome amplification. Nat Commun. 2016 Oct 31;7:13227. doi: 10.1038/ncomms13227. PMID 27796307
- [Result] Jiang Y, Hsieh J. HDAC3 controls gap 2/mitosis progression in adult neural stem/progenitor cells by regulating CDK1 levels. Proc Natl Acad Sci U S A. 2014 Sep 16;111(37):13541-6. doi: 10.1073/pnas.1411939111. Epub 2014 Aug 26. PMID 25161285
- [Derived] Li G, Ma X, Zhao H, Fan J, Liu T, Luo Y, Guo Y. Long non-coding RNA H19 promotes leukocyte inflammation in ischemic stroke by targeting the miR-29b/C1QTNF6 axis. CNS Neurosci Ther. 2022 Jun;28(6):953-963. doi: 10.1111/cns.13829. Epub 2022 Mar 24. PMID 35322553